CLINICAL TRIAL: NCT01173588
Title: Effect of Yogurt Added With Bifidobacteria and Soluble Fiber on Bowel Function: A Randomized, Double-blind, Longitudinal Controlled Study in Mexican Adult.
Brief Title: Effect of Yogurt Added With Bifidobacteria and Soluble Fiber on Bowel Function.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Lala (Industry)
Collaborators: Cindetec (Other)
Responsible Party: Jorge Luis Rosado Loría, Universidad autonoma de queretaro
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEE-001-2007
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: bowel function; functional foods
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yogurt+fiber+probiotic (Experimental): Yogurt YBF was added with 1.5 g inulin/100 g and ≥5 x 107 CFU of bifidobacterium/mL
  Interventions: Other: yogurt added with bifidobacteria and soluble fiber (YBF)
- regular yogurt (Placebo Comparator): yogurt YR had no additional fiber or bifidobacterium
  Interventions: Other: yogurt added with bifidobacteria and soluble fiber (YBF)

INTERVENTIONS:
Other: yogurt added with bifidobacteria and soluble fiber (YBF) — Yogurt in YBF was added with 1.5 g inulin/100 g and ≥5 x 107 CFU of bifidobacterium/mL
  Other Names: yogurt LALA Vive; Yogurt LALA regular

SUMMARY:
The aim of this study was to evaluate the effect of the consumption of yogurt added with bifidobacteria and soluble fiber on gastrointestinal function of healthy adults. A product as herein described is expected to improve gastrointestinal function and maintain the intestinal microflora balance of healthy subjects and perhaps of patients with altered bowel functions.

DETAILED DESCRIPTION:
The use of probiotics and prebiotics has become popular in human nutrition and food product development. The most common probiotics are Lactobacillus and Bifidobacterium species. Bifidobacteria spp are dominant in the intestinal microflora and are considered to be beneficial to the host, for this reason research efforts have focused on increasing their proportion in the intestinal microflora through oral administration of mixtures containing bifidobacteria or oral supplementation with prebiotics. An important limitation for the effectiveness of oral probiotics is that they might be destroyed during digestion in the gastrointestinal tract therefore and adequate vehicle could improve its potential benefits. Yogurt is a suitable vehicle for the administration of bifidobacteria, due to its physicochemical properties, such as pH and nutrients content, as well as the organoleptic properties that contribute to its increasing consumption. Thus simultaneous administration of probiotics and prebiotics in a suitable vehicle could act synergistically and may have potential for improving gut health. Few clinical trials have been performed using prebiotics and probiotics. The aim of this study was to evaluate the effect of the consumption of yogurt added with bifidobacteria and soluble fiber on gastrointestinal function of healthy adults. A product as herein described is expected to improve gastrointestinal function and maintain the intestinal microflora balance of healthy subjects and perhaps of patients with altered bowel functions.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years,
* be free of known gastrointestinal diseases,
* desist of consuming prebiotic and/or probiotic-containing foods or dietary supplements during the entire duration of the study,
* agree to avoid any medication that produced changes in gastrointestinal function, diarrhea or constipation until completion of the study,
* be willing to complete all necessary study questionnaires,
* accept voluntary participation and sign a written informed consent before inclusion in the study.

Exclusion Criteria:

* subjects receiving any kind of treatment that may had altered bowel function;
* intake of laxatives,
* a concomitant sever gastrointestinal disease;
* that were consuming probiotics and/or prebiotics-containing foods or dietary supplements within the two previous weeks;
* subjects were also excluded if they had received any antimicrobial medication during the previous 2 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2007-06; Primary Completion 2007-12 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Stools Frequency | 0, 1, 2, 3, 4, 5 weeks
  Stools frequency was reported daily as follows: 0: zero 1= once, 2= twice, 3=three times, 4= four or more times

SECONDARY OUTCOMES:
Consistency of stools | 0, 1, 2, 3, 4, 5 weeks
  Consistency of stools was scored according to the following scale: 1= watery and liquid, 2= soft and unformed, 3= soft and formed, and 4= hard and dry.
Difficulty of defecation | 0,1,2,3,4,5
  Difficulty of defecation was evaluated as 1= very easy, 2= easy, 3= hard, 4= very hard.
Abdominal distension | 0,1,2,3,4,5
  Abdominal distension was evaluated as 1= no symptoms, 2= slight symptoms that did not influence daily activities, 3= moderate symptoms that could influence daily activities, 4= severe symptoms that affected daily activities.
Flatulence | 0,1,2,3,4,5
  Flatulence was evaluated as 1= no symptoms, 2= slight symptoms that did not influence daily activities, 3= moderate symptoms that could influence daily activities, 4= severe symptoms that affected daily activities.
Abdominal pain | 0,1,2,3,4,5 weeks
  Abdominal pain was evaluated as 1= no symptoms, 2= slight symptoms that did not influence daily activities, 3= moderate symptoms that could influence daily activities, 4= severe symptoms that affected daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge JL Rosado, PhD, Principal Investigator — UAQ
Locations (1):
- Cindetec, Querétaro City, Querétaro, Mexico